CLINICAL TRIAL: NCT01200511
Title: A Prospective Pilot Clinical Study of the AcrySof® IQ ReSTOR® Multifocal Toric IOL
Brief Title: Pilot Study of AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M09-052
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-03

CONDITIONS: Cataract
Keywords: intraocular lens; multifocal; toric
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReSTOR +3.0 (Experimental): AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism, bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL — Multifocal IOL with extended secondary focal point and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Other Names: Models SND1T3, SND1T4, SND1T5

SUMMARY:
The purpose of this study is to describe visual outcomes, in particular spherical equivalent by manifest refraction and visual acuity across a range of distances, 6 months post implantation of the AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL in adult patients with corneal astigmatism. Additionally, patient reported outcomes will be assessed.

DETAILED DESCRIPTION:
Each subject completed a preoperative examination of both eyes, implantation of IOL at the operative visit for each eye, and up to 5 postoperative visits (each eye examined at Day 1-2, with binocular visits at Month 1, Month 3, and Month 6 after the second implantation). The second implantation generally occurred within 30 days of the first.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Require cataract extraction followed by posterior IOL implantation or eligible for refractive lens exchange (RLE) in both eyes;
* Able to undergo second eye surgery within one month (30 days) of first eye surgery;
* Able to attend postoperative examinations per protocol schedule;
* Qualify for a AcrySof IQ Toric IOL in both eyes;
* Preoperative astigmatism of ≥0.75 to ≤2.5 diopters (D) in both eyes;
* Residual refractive cylinder of ≤0.5 D in both eyes;
* Good ocular health;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Planned multiple procedures, including LRI, during cataract/IOL implantation surgery;
* Amblyopia;
* Previous corneal surgery;
* Clinically significant corneal endothelial dystrophy;
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.);
* History of retinal detachment;
* Pregnant or planning to become pregnant during course of study;
* Other protocol-defined exclusion criteria may apply.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brand Lead, Surgical, Global Medical Affairs, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 investigational sites located in Germany (2), Venezuela (2), and Spain (1).
Pre-assignment Details: This reporting population includes all enrolled subjects.
Groups:
- ReSTOR +3.0 Toric: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism, bilateral implantation
Period: Overall Study
Arm/Group | ReSTOR +3.0 Toric
Started | 49
Completed | 44
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all patients receiving IOL implantation in both eyes that completed the study.
Arm/Group | ReSTOR +3.0 Toric
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.52 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Visual Acuity Across a Range of Distances at Month 6
Description: Visual acuity (VA) was tested binocularly (both eyes together) unaided across a range of distances under well-lit conditions using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Month 6 from second eye implantation
Population: This analysis population includes all subjects receiving IOL implantation in both eyes with data at visit.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR +3.0 Toric
Number analyzed (Participants) | 42
logMAR
  Far distance 4 meters (m) | 0.05 (0.10)
  Intermediate 70 centimeters (cm) | 0.15 (0.13)
  Intermediate 60 cm | 0.09 (0.11)
  Intermediate 50 cm | 0.05 (0.09)
  Near 40 cm | 0.07 (0.09)
  Near - preferred | 0.04 (0.08)

2. Primary Outcome: Best Corrected Visual Acuity (BCVA) Across a Range of Distances at Month 6
Description: VA was tested binocularly with correction in place if needed across a range of distances under well-lit conditions using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Month 6 from second eye implantation
Population: This analysis population includes all subjects receiving IOL implantation in both eyes with data at visit.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR +3.0 Toric
Number analyzed (Participants) | 42
logMAR
  Far distance 4 m | 0.00 (0.06)
  Intermediate 70 cm | 0.19 (0.14)
  Intermediate 60 cm | 0.14 (0.14)
  Intermediate 50 cm | 0.06 (0.10)
  Near 40 cm | 0.04 (0.07)
  Near - preferred distance | 0.05 (0.08)

3. Primary Outcome: Proportion of Subjects That Achieved Spherical Equivalent Within ± 0.5D, ± 0.75D, and ± 1.0D at Month 6
Description: Manifest refraction was performed under well-lit conditions using an ETDRS chart. The subject was manually refracted to his/her best correction by an outcomes assessor using a phoropter or trial lenses. Manifest refraction was performed for each eye. Proportion of subjects that achieved spherical equivalent within ± 0.5D/ ± 0.75D/ ± 1.0D at Month 6 is reported as percentage of subjects.
Time Frame: Month 6 from second eye implantation
Population: This analysis population includes all subjects receiving IOL implantation in both eyes with data at visit.
Measure: Number; unit: percentage of participants
Arm/Group | ReSTOR +3.0 Toric
Number analyzed (Participants) | 44
percentage of participants
  ± 0.5D | 84.5
  ± 0.75D | 92.9
  ±1.0D | 95.2

4. Secondary Outcome: Patient Reported Outcomes at Month 6
Description: The Visual Task Difficulty Assessment (VISTAS) questionnaire was completed by the subject to assess difficulty in completing everyday tasks that depend on good vision. Distance specific tasks were rated (without / with corrective aids) using a 1 to 5 point scale, where 1 = no difficulty; 2 = minor difficulty; 3 = moderate difficulty; 4 = major difficulty; 5 = cannot accomplish. Individual scores for each task were averaged to obtain the overall score for each vision type/function. Near vision was defined as less than 50 cm; intermediate vision as 50 cm to 1 m; extended intermediate vision as 90 cm to 4 m; and distant vision as more than 4 m.
Time Frame: Month 6 from second eye implantation
Population: This analysis population includes all subjects receiving IOL implantation in both eyes with data at visit. A subject may have responded with and without.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ReSTOR +3.0 Toric/Without: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism, bilateral implantation, without corrective aids
- ReSTOR +3.0 Toric/With: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism, bilateral implantation, with corrective aids if needed
Arm/Group | ReSTOR +3.0 Toric/Without | ReSTOR +3.0 Toric/With
Number analyzed (Participants) | 44 | 44
units on a scale
  Near function scale score: number analyzed (Participants) | 39 | 5
  Near function scale score | 1.72 (0.65) | 1.65 (0.60)
  Intermediate function scale score: number analyzed (Participants) | 39 | 6
  Intermediate function scale score | 1.49 (0.59) | 1.21 (0.51)
  Extended intermediate function scale score: number analyzed (Participants) | 39 | 7
  Extended intermediate function scale score | 1.24 (0.38) | 1.20 (0.37)

ADVERSE EVENTS:
Time Frame: An Adverse Event (AE) was defined as any untoward medical occurrence in a subject, user, or other persons regardless of causal relationship.
Description: This analysis population includes all enrolled subjects that underwent surgery independent of IOL implantation.
Arm/Group | ReSTOR +3.0 Toric
Serious Adverse Events (participants affected / at risk) | 7/49
Other Adverse Events (participants affected / at risk) | 3/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR +3.0 Toric (N=49)
Macular oedema (Eye disorders) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 1
Device dislocation (General disorders) | 3
Intraocular pressure test abnormal (Investigations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Intraocular Lens Repositioning (Surgical and medical procedures) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ReSTOR +3.0 Toric (N=49)
Posterior capsule opacification (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.